CLINICAL TRIAL: NCT02898909
Title: Comparison of Two Fragmentation Modalities in Femtosecond Laser-assisted Cataract Surgery
Acronym: SLICES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Major inclusion difficulties
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JFO_2015_44
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Cataract
Keywords: femtosecond laser-assisted cataract surgery; nuclear lens fragmentation
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 16 pieces fragmentation (Experimental)
  Interventions: Device: nuclear lens fragmentation in 16 pieces
- 8 pieces fragmentation (Active Comparator)
  Interventions: Device: nuclear lens fragmentation in 8 pieces

INTERVENTIONS:
Device: nuclear lens fragmentation in 8 pieces
  Arms: 8 pieces fragmentation
Device: nuclear lens fragmentation in 16 pieces
  Arms: 16 pieces fragmentation

SUMMARY:
Femtosecond laser-assisted cataract surgery consists in nuclear lens fragmentation, followed by ultrasound phacoemulsification of nuclear lens, which is then removed.

It can be assumed that fragmenting the nuclear lens in more pieces could facilitate the post-laser ultrasound phacoemulsification to extract the lens, with a lesser amount of ultrasonic energy.

The decrease of ultrasonic energy delivered during cataract surgery is beneficial to the patient because it optimizes the vitality of corneal endothelial cells, which ensure corneal transparency.

ELIGIBILITY:
Inclusion Criteria:

* patient aged ≥ 18 years old
* first Femtosecond Laser-assisted Cataract Surgery scheduled
* cataract density ≥ 3 according to the lens opacities classification system (LOCS)

Exclusion Criteria:

* corneal guttata, uncontrolled glaucoma
* shallow depth of anterior chamber
* patient's refusal to participate in the study
* pregnant or breast feeding patient
* patient under legal protection
* no health coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
energy delivered for lens nucleus aspiration during phacoemulsification | approximatively 15 minutes
  ultrasound power delivered (measured in Hertz)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc FEBBRARO, MD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation Opthalmologique A de Rothschild, Paris, France